CLINICAL TRIAL: NCT00064194
Title: A Double-Blind, Placebo-Controlled, Randomized Study Of Combination Vitamin E, Selenium And Soy Protein Product In Subjects With High Grade Prostatic Intraepithelial Neoplasia
Brief Title: Vitamin E, Selenium, and Soy Protein in Preventing Cancer in Patients With High-Grade Prostate Neoplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Masking: Triple | Purpose: Prevention
Other Study IDs: PRP1; CAN-NCIC-PRP1 (Other: PDQ); CDR0000310096 (Other: PDQ)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Precancerous/Nonmalignant Condition; Prostate Cancer
Keywords: prostate cancer; high grade prostatic intraepithelial neoplasia
MeSH Terms: conditions — Precancerous Conditions; Prostatic Neoplasms | interventions — Selenium; Soybean Proteins; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: selenium
Dietary Supplement: soy protein isolate
Dietary Supplement: vitamin E

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain substances to try to prevent the development or recurrence of cancer. Vitamin E, selenium, and soy protein may be effective in preventing the development of prostate cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of combining vitamin E, selenium, and soy protein in preventing prostate cancer in patients who have high-grade prostate neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether nutritional supplementation with soy protein isolate, vitamin E, and selenium can delay the time to development of invasive prostate cancer (disease-free survival) in patients with high-grade prostatic intraepithelial neoplasia.
* Determine the effect of this supplementation on intermediate endpoints that may reflect a lessened risk of invasive prostate cancer (e.g., serum PSA levels, hormone levels, lycopene, malondialdehyde, vitamin E, and reduced thiol groups) in these patients.
* Determine the safety of this supplementation in these patients.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral vitamin E, oral selenium, and oral soy protein isolate twice daily.
* Arm II: Patients receive oral placebo twice daily. In both arms, treatment continues for 3 years in the absence of invasive prostate cancer (demonstrated on biopsy) or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 306 patients (153 per treatment arm) will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-grade prostatic intraepithelial neoplasia (HGPIN)

  * No evidence of invasive prostate cancer by at least 2 biopsies within the past 18 months
  * At least 1 biopsy must show evidence of HGPIN within the past 6 months
* No prior invasive prostate cancer

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Not specified

Life expectancy

* More than 5 years

Hematopoietic

* Platelet count at least 75,000/mm^3
* No coagulopathies

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* PT (INR) no greater than 1.5 times ULN
* PTT no greater than 1.5 times ULN
* No hepatic insufficiencies

Renal

* Creatinine no greater than 2 times ULN
* No renal insufficiencies

Other

* No prior nonmelanoma skin cancer (e.g., squamous cell or basal cell carcinoma)
* No other malignancy within the past 5 years except superficial bladder cancer
* No known bowel malabsorption
* No dietary behavior (e.g., morbid obesity or eating disorders) that would limit adherence to study therapy
* No major illness, including psychiatric illness, that would preclude study compliance and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* More than 3 months since prior androgen therapy
* More than 3 months since prior hormonal therapy for benign prostatic hyperplasia (e.g., finasteride)
* No concurrent finasteride
* No concurrent androgen therapy

Radiotherapy

* More than 2 years since prior radiotherapy to the pelvic region

Surgery

* Not specified

Other

* More than 2 weeks since prior supplemental vitamin E or selenium
* No other concurrent vitamin E (greater than 100 IU/day), selenium, or soy protein isolate (more than 2 servings/week)
* No other concurrent treatment for high-grade prostatic intraepithelial neoplasia

Max Age: 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2001-11-28 (Actual); Primary Completion 2008-04-30 (Actual); Study Completion 2008-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Fleshner, Study Chair — Princess Margaret Hospital, Canada
Locations (3):
- Canada (3):
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fleshner NE, Kapusta L, Donnelly B, Tanguay S, Chin J, Hersey K, Farley A, Jansz K, Siemens DR, Trpkov K, Lacombe L, Gleave M, Tu D, Parulekar WR. Progression from high-grade prostatic intraepithelial neoplasia to cancer: a randomized trial of combination vitamin-E, soy, and selenium. J Clin Oncol. 2011 Jun 10;29(17):2386-90. doi: 10.1200/JCO.2010.32.0994. Epub 2011 May 2. PMID 21537051